CLINICAL TRIAL: NCT01978834
Title: Age Dependend Diagnostic Thresholds for Osteoporosis Bindex Ultrasonometer
Status: Completed | Type: Observational
Sponsor: Bone Index Finland Ltd (Industry)
Collaborators: HealthPartners Institute (Other)
Responsible Party: Sponsor
Other Study IDs: Bind02; BoneIndex02 (Other: Bone Index Finland Ltd.)
Record Dates: First submitted 2013-10-28; First posted 2013-11-08 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Osteoporosis
Keywords: Osteoporosis, diagnosis, ultrasound
MeSH Terms: conditions — Osteoporosis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is designed for clinical validation of the novel ultrasound device (Bindex®, Bone Index Finland Ltd.). In a preliminary study technique has been validated in Finnish elderly woman population with 285 healthy and 56 osteoporotic subjects (n = 341 in total). Significant and good correlation was observed between Density Index (DI) determined with Bindex and femoral bone mineral density determined with DXA (r = 0.65 - 0.70). In addition, with determination of 90% sensitivity and specificity thresholds, significant number (65-75%) of patients could be diagnosed without additional verification with DXA.

First, the thresholds for DI will be determined by measuring 70 osteoporotic and 70 healthy patients (n = 140) with Bindex and DXA within four decades of age; age 50 to 59 years, age 60 to 69 years, age 70 to 79 years, and age 80 to 89 years. The feasibility of DI for diagnostics of osteoporosis and evaluation of bone mineral density (BMD) will be assessed. The thresholds for the BMD estimate obtained with DI will be determined for osteoporotic and non-osteoporotic patients. For fracture risk assessment, DI measurements are used to predict the outcome of currently available fracture risk assessment tools.

1. To investigate optimal configuration of ultrasound parameters and patient characteristics for prediction of proximal femur and lumbar spine BMD for women in each four decades of age; 50 to 59 years, 60 to 69 years, 70 to 79 years, and 80-89 years.
2. To develop national diagnostic thresholds for DI in prediction of osteoporosis status with a reference female population (American-Caucasian) in each four decades of age; 50 to 59 years, 60 to 69 years, 70 to 79 years, and 80-89 years.

DETAILED DESCRIPTION:
Data will be stored by Park Nicollet Institute. Only data listed below will be given to the research team at Bindex for analyses.

The data for determination of diagnostic threshold for DI in North American population will be analyzed by Bone Index Finland. The data will include following parameters:

* Age in years
* Weight
* Height
* Cortical thickness values at each location
* Density Index values
* Raw data on ultrasound signals.
* DXA measurement data
* Identification code (Uniquely created identification code given to a subject, does not carry any information on subject but enables tracing if needed.)
* Data from Appendix A, excluding patient name and medical record number

Risk factors will be collected in a separate questionnaire (Appendix A).

1. Name
2. Medical Record Number
3. Weight (kg)
4. Height (cm)
5. Chair Stand test Can do easily; can do only with difficulty; cannot do

   Risk Factors:
6. Previous fracture (Skeletal site, age at which fracture occured)
7. Parent fractured hip (Yes, No)
8. Current smoking (Yes, No)
9. Glucocorticoid Use (Yes, No)
10. Rheumatoid arthritis (Yes, No)
11. Alcohol 3 or more units per day (Yes, No)
12. Osteoporosis medication, type (e.g. alendronate, bisphosphonates), start- and end-date (Within the past five years)

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Age 50 to 89 years

Exclusion Criteria:

* Those who have opted out of being contacted for research on their general Park Nicollet clinic consent will not be recruited by mail
* Inability to sign consent form due to cognitive impairment. Those with dementia (ICD-9 diagnosis codes 331.0, 294.1, 294.10, 294.11, or 294.8) will excluded from mailed recruitment
* Measurement of hip BMD is not feasible (for example, those who have had bilateral hip replacement surgeries or who cannot have central DXA because of their body weight)
* Open leg or arm wounds at sites where ultrasound measurements are supposed to be taken, precluding such measurements

Ages: 50 Years to 89 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female (American-Caucasian)
Sampling Method: Non-Probability Sample
Enrollment: 560 (Actual)
Dates: Start 2013-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Thresholds for Bindex in Osteoporosis Diagnostics | 1 year
  Diagnostics thresholds for DI parameter for Osteoporosis within four decades of age; age 50 to 59 years, age 60 to 69 years, age 70 to 79 years, and age 80 to 89 years.

CONTACTS AND LOCATIONS:
Overall Officials: John T Schousboe, MD, PhD, Principal Investigator — HealthPartners Institute; Janne P Karjalainen, PhD, Study Director — Bone Index Finland Ltd; Ossi Riekkinen, PhD, Study Director — Bone Index Finland Ltd
Locations (1):
- Park Nicollet Institute, Minneapolis, Minnesota, United States